CLINICAL TRIAL: NCT04676126
Title: Augmented Macular Pigment Supplement and Pericentral Visual Function: a Randomized Controlled Trial
Brief Title: Augmented Macular Pigment-containing Nutraceutical and Central Visual Function
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB records show administrative closure on 12/16/21. No subjects enrolled.
Sponsor: University of the Incarnate Word (Other)
Collaborators: Guardion Health Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-11-005
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma; Glaucoma Eye; Glaucoma, Open-Angle
Keywords: Lumega-Z; Macular Pigment; Macular Pigment Optical Density; Contrast Sensitivity; Humphrey Visual Field 10-2; Dermal Carotenoid; MapcatSF; Veggie Meter; Vector Vision; Pericentral Visual Field
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — dorzolamide; brinzolamide

STUDY DESIGN:
Intervention Model Description: This is a prospective double-masked, randomized controlled study which compares pre- supplementation macular pigment optical density, contrast sensitivity, dermal carotenoid levels, and visual field status to post-supplement measurements of the same.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A remotely located Guardion Health Sciences designee will utilize a computer-generated random number table to assign patients to placebo or experimental group. Subjects will have the supplement/placebo delivered to their homes in identical (except lot number) packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects in the experimental arm will consume 1.5 Tbsp (22.2 mL) of a commercial macular pigment-containing medical food (liquid) once per day and use a carbonic anhydrase inhibitor topical eye drop (2% dorzolamide ophthalmic solution) three times per day in both eyes for 3 months.
  Interventions: Dietary Supplement: Lumega-Z; Drug: Dorzolamide Hcl 2% Oph Soln
- Placebo (Placebo Comparator): Subjects in the placebo arm will consume 1.5 Tbsp (22.2 mL) of a placebo liquid which resembles the commercial macular pigment-containing medical food (liquid) in taste once per day and use a lubricating eye drop (0.5% sodium + 0.9% glycerin ophthalmic solution) three times per day in both eyes for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lumega-Z — Medical food which contains lutein, zeaxanthin, and meso-zeaxanthin
  Arms: Experimental
Drug: Dorzolamide Hcl 2% Oph Soln — Topical carbonic anhydrase inhibitor
  Other Names: Azopt
  Arms: Experimental
Other: Placebo — Specially formulated non macular pigment-containing formulation which tastes similar to the commercial medical food being evaluated in this study
  Arms: Placebo

SUMMARY:
The purpose of this study is to prospectively analyze changes in macular pigment optical density and dermal carotenoid levels as they relate to visual field function in patients prescribed a macular pigment-containing medical food (Lumega-Z), in combination with a topical carbonic anhydrase inhibitor.

DETAILED DESCRIPTION:
This is a prospective double-masked, randomized controlled trial which evaluates central visual field function as it relates to macular pigment optical density, contrast sensitivity, and dermal carotenoid levels in the presence of a commercial macular pigment-containing medical food (Lumega-Z). Participants will be randomized to twelve weeks of supplement + dorzolamide or twelve weeks of placebo. All packaging of supplement and dorzolamide and the placebo will be identical and distributed by a third party. Both subjects and the investigators examining patients will be masked to placebo and experimental group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Glaucoma diagnosis (H40. *) with abnormal visual field as measured by 30-2 Humphrey Perimetry (mean deviation < -2.00)
* Adequate IOP control (IOP > 7 mmHg and < 22 mmHg) by medical or surgical means measured by Goldman Applanation Tonometry for at least 3 months
* Visual field progression - decrease (more negative) in MD by 1.00 dB or more when compared to prior HVF)
* Refractive error ≤ 10 diopters and astigmatism ≤ 3 diopters

Exclusion Criteria:

* BCVA worse than 20/200
* Pt Is unable to tolerate MPOD, CS, dermal carotenoid measurement-taking procedures
* Loss of IOP control requires surgical intervention
* Patient already taking AREDS formula oral supplement
* Patient taking medication or dietary supplements that may interact with LM ingredients
* History of photosensitive epilepsy
* History of penetrating ocular trauma or vitrectomy
* History of ocular or orbital radiation therapy or is currently receiving chemotherapy
* Women who are nursing, pregnant, or are planning pregnancy
* Has a known adverse reaction (including sulfa allergy) and/or sensitivity to the study supplement or its ingredients including: N-acetyl-cysteine, acetyl-L-carnitine, L-taurine, quercetin, Co-enzyme Q-10, lutein, meso zeaxanthin, zeaxanthin, astazanthin, lycopene, alpha-lipoic acid.
* Currently enrolled in an investigational drug study or has used an investigational drug within 30 days prior to recruitment.
* Is planning on having ocular surgery at any time throughout the study duration, or had ocular surgery < 3 months before enrollment
* Native lens opacity ≥ grade 3 on ARLNS standard photograph
* Blue light filter intraocular lens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Pericentral Visual Function | 3 Months
  Mean deviation and pattern standard deviation of 10-2 Humphrey visual field

SECONDARY OUTCOMES:
Macular Pigment Optical Density | Monthly for 3 months
  Macular Pigment Optical Density measured by Mapcat SF
Dermal Carotenoid Levels | Monthly for 3 months
  Measured by Veggie Meter
Contrast Sensitivity | Monthly for 3 months
  Measured by Vector Vision CSV-2000

CONTACTS AND LOCATIONS:
Overall Officials: Grant T Slagle, DO, Principal Investigator — Sponsel Foundation
Locations (1):
- Ophtalmology Clinic of William E Sponsel, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researches.

REFERENCES:
- [Background] Bone RA, Davey PG, Roman BO, Evans DW. Efficacy of Commercially Available Nutritional Supplements: Analysis of Serum Uptake, Macular Pigment Optical Density and Visual Functional Response. Nutrients. 2020 May 6;12(5):1321. doi: 10.3390/nu12051321. PMID 32384663
- [Background] Ma L, Liu R, Du JH, Liu T, Wu SS, Liu XH. Lutein, Zeaxanthin and Meso-zeaxanthin Supplementation Associated with Macular Pigment Optical Density. Nutrients. 2016 Jul 12;8(7):426. doi: 10.3390/nu8070426. PMID 27420092
- [Background] Power R, Coen RF, Beatty S, Mulcahy R, Moran R, Stack J, Howard AN, Nolan JM. Supplemental Retinal Carotenoids Enhance Memory in Healthy Individuals with Low Levels of Macular Pigment in A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Alzheimers Dis. 2018;61(3):947-961. doi: 10.3233/JAD-170713. PMID 29332050
- [Background] Jahns L, Johnson LK, Mayne ST, Cartmel B, Picklo MJ Sr, Ermakov IV, Gellermann W, Whigham LD. Skin and plasma carotenoid response to a provided intervention diet high in vegetables and fruit: uptake and depletion kinetics. Am J Clin Nutr. 2014 Sep;100(3):930-7. doi: 10.3945/ajcn.114.086900. Epub 2014 Jul 9. PMID 25008856
- [Background] Jahns L, Johnson LK, Conrad Z, Bukowski M, Raatz SK, Jilcott Pitts S, Wang Y, Ermakov IV, Gellermann W. Concurrent validity of skin carotenoid status as a concentration biomarker of vegetable and fruit intake compared to multiple 24-h recalls and plasma carotenoid concentrations across one year: a cohort study. Nutr J. 2019 Nov 21;18(1):78. doi: 10.1186/s12937-019-0500-0. PMID 31752882
- [Background] Conrady CD, Bell JP, Besch BM, Gorusupudi A, Farnsworth K, Ermakov I, Sharifzadeh M, Ermakova M, Gellermann W, Bernstein PS. Correlations Between Macular, Skin, and Serum Carotenoids. Invest Ophthalmol Vis Sci. 2017 Jul 1;58(9):3616-3627. doi: 10.1167/iovs.17-21818. PMID 28728169
- [Background] Ermakov IV, Gellermann W. Dermal carotenoid measurements via pressure mediated reflection spectroscopy. J Biophotonics. 2012 Jul;5(7):559-70. doi: 10.1002/jbio.201100122. Epub 2012 Feb 13. PMID 22331637
- [Background] Sponsel WE, Harrison J, Elliott WR, Trigo Y, Kavanagh J, Harris A. Dorzolamide hydrochloride and visual function in normal eyes. Am J Ophthalmol. 1997 Jun;123(6):759-66. doi: 10.1016/s0002-9394(14)71124-9. PMID 9535619
- [Background] Bone RA, Landrum JT, Hime GW, Cains A, Zamor J. Stereochemistry of the human macular carotenoids. Invest Ophthalmol Vis Sci. 1993 May;34(6):2033-40. PMID 8491553
- [Background] Britton G. Structure and properties of carotenoids in relation to function. FASEB J. 1995 Dec;9(15):1551-8. PMID 8529834
- [Background] Age-Related Eye Disease Study 2 (AREDS2) Research Group; Chew EY, Clemons TE, Sangiovanni JP, Danis RP, Ferris FL 3rd, Elman MJ, Antoszyk AN, Ruby AJ, Orth D, Bressler SB, Fish GE, Hubbard GB, Klein ML, Chandra SR, Blodi BA, Domalpally A, Friberg T, Wong WT, Rosenfeld PJ, Agron E, Toth CA, Bernstein PS, Sperduto RD. Secondary analyses of the effects of lutein/zeaxanthin on age-related macular degeneration progression: AREDS2 report No. 3. JAMA Ophthalmol. 2014 Feb;132(2):142-9. doi: 10.1001/jamaophthalmol.2013.7376. PMID 24310343
- [Background] Aronow ME, Chew EY. Age-related Eye Disease Study 2: perspectives, recommendations, and unanswered questions. Curr Opin Ophthalmol. 2014 May;25(3):186-90. doi: 10.1097/ICU.0000000000000046. PMID 24614146
- [Background] Akuffo KO, Beatty S, Peto T, Stack J, Stringham J, Kelly D, Leung I, Corcoran L, Nolan JM. The Impact of Supplemental Antioxidants on Visual Function in Nonadvanced Age-Related Macular Degeneration: A Head-to-Head Randomized Clinical Trial. Invest Ophthalmol Vis Sci. 2017 Oct 1;58(12):5347-5360. doi: 10.1167/iovs.16-21192. PMID 29053808
- [Background] Nakano Y, Hirooka K, Chiba Y, Ueno M, Ojima D, Hossain MR, Takahashi H, Yamamoto T, Kiuchi Y. Retinal ganglion cell loss in kinesin-1 cargo Alcadein alpha deficient mice. Cell Death Dis. 2020 Mar 3;11(3):166. doi: 10.1038/s41419-020-2363-x. PMID 32127528
- [Background] Quigley HA. Glaucoma. Lancet. 2011 Apr 16;377(9774):1367-77. doi: 10.1016/S0140-6736(10)61423-7. Epub 2011 Mar 30. PMID 21453963
- [Background] Knox DL, Eagle RC Jr, Green WR. Optic nerve hydropic axonal degeneration and blocked retrograde axoplasmic transport: histopathologic features in human high-pressure secondary glaucoma. Arch Ophthalmol. 2007 Mar;125(3):347-53. doi: 10.1001/archopht.125.3.347. PMID 17353405
- [Background] Tsai T, Reinehr S, Maliha AM, Joachim SC. Immune Mediated Degeneration and Possible Protection in Glaucoma. Front Neurosci. 2019 Sep 2;13:931. doi: 10.3389/fnins.2019.00931. eCollection 2019. PMID 31543759
- [Background] Pinazo-Duran MD, Zanon-Moreno V, Gallego-Pinazo R, Garcia-Medina JJ. Oxidative stress and mitochondrial failure in the pathogenesis of glaucoma neurodegeneration. Prog Brain Res. 2015;220:127-53. doi: 10.1016/bs.pbr.2015.06.001. Epub 2015 Sep 8. PMID 26497788
- [Background] Greco A, Rizzo MI, De Virgilio A, Gallo A, Fusconi M, de Vincentiis M. Emerging Concepts in Glaucoma and Review of the Literature. Am J Med. 2016 Sep;129(9):1000.e7-1000.e13. doi: 10.1016/j.amjmed.2016.03.038. Epub 2016 Apr 26. PMID 27125182
- [Background] Wax MB. The case for autoimmunity in glaucoma. Exp Eye Res. 2011 Aug;93(2):187-90. doi: 10.1016/j.exer.2010.08.016. Epub 2010 Aug 27. PMID 20801114
- [Background] Foote CS, Chang YC, Denny RW. Chemistry of singlet oxygen. X. Carotenoid quenching parallels biological protection. J Am Chem Soc. 1970 Aug 26;92(17):5216-8. doi: 10.1021/ja00720a036. No abstract available. PMID 5432666
- [Background] Mayne ST, Cartmel B, Scarmo S, Jahns L, Ermakov IV, Gellermann W. Resonance Raman spectroscopic evaluation of skin carotenoids as a biomarker of carotenoid status for human studies. Arch Biochem Biophys. 2013 Nov 15;539(2):163-70. doi: 10.1016/j.abb.2013.06.007. Epub 2013 Jun 30. PMID 23823930
- [Background] Obana A, Tanito M, Gohto Y, Okazaki S, Gellermann W, Bernstein PS. Changes in Macular Pigment Optical Density and Serum Lutein Concentration in Japanese Subjects Taking Two Different Lutein Supplements. PLoS One. 2015 Oct 9;10(10):e0139257. doi: 10.1371/journal.pone.0139257. eCollection 2015. PMID 26451726
- [Background] Schmidl D, Schmetterer L, Garhofer G, Popa-Cherecheanu A. Pharmacotherapy of glaucoma. J Ocul Pharmacol Ther. 2015 Mar;31(2):63-77. doi: 10.1089/jop.2014.0067. Epub 2015 Jan 14. PMID 25587905
- [Background] Eysteinsson T, Gudmundsdottir H, Hardarson AO, Berrino E, Selleri S, Supuran CT, Carta F. Carbonic Anhydrase Inhibitors of Different Structures Dilate Pre-Contracted Porcine Retinal Arteries. Int J Mol Sci. 2019 Jan 22;20(3):467. doi: 10.3390/ijms20030467. PMID 30678227
- [Background] Remky A, Weber A, Arend O, Sponsel WE. Topical dorzolamide increases pericentral visual function in age-related maculopathy: pilot study findings with short-wavelength automated perimetry. Acta Ophthalmol Scand. 2005 Apr;83(2):154-60. doi: 10.1111/j.1600-0420.2005.00406.x. PMID 15799725
- [Background] Hammond BR Jr, Fuld K. Interocular differences in macular pigment density. Invest Ophthalmol Vis Sci. 1992 Feb;33(2):350-5. PMID 1740365
- [Background] Chew EY, Clemons TE, Agron E, Sperduto RD, Sangiovanni JP, Kurinij N, Davis MD; Age-Related Eye Disease Study Research Group. Long-term effects of vitamins C and E, beta-carotene, and zinc on age-related macular degeneration: AREDS report no. 35. Ophthalmology. 2013 Aug;120(8):1604-11.e4. doi: 10.1016/j.ophtha.2013.01.021. Epub 2013 Apr 10. PMID 23582353
- [Background] Katz LJ, Simmons ST, Craven ER. Efficacy and safety of brimonidine and dorzolamide for intraocular pressure lowering in glaucoma and ocular hypertension. Curr Med Res Opin. 2007 Dec;23(12):2971-83. doi: 10.1185/030079907X242476. PMID 17949534
- [Background] Padmanaban V, Inati S, Ksendzovsky A, Zaghloul K. Clinical advances in photosensitive epilepsy. Brain Res. 2019 Jan 15;1703:18-25. doi: 10.1016/j.brainres.2018.07.025. Epub 2018 Aug 1. PMID 30076791

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04676126/Prot_SAP_002.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04676126/ICF_003.pdf